CLINICAL TRIAL: NCT02401542
Title: A Dose Escalation, Expansion Study of Vofatamab (B-701) Alone, Plus Docetaxel, or Versus Docetaxel in Subjects With Locally Advanced or Metastatic Urothelial Cell Carcinoma Who Have Relapsed After, or Are Refractory to Standard Therapy
Brief Title: Dose Escalation, Expansion Study of Vofatamab (B-701) in Treatment of Locally Advanced or Metastatic Urothelial Cell Carcinoma
Acronym: FIERCE-21
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: program has been put on hold by the sponsor
Sponsor: Rainier Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-701-U21; 2017-001319-36 (EudraCT Number)
Record Dates: First submitted 2015-03-16; First posted 2015-03-30 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Locally Advanced or Metastatic Urothelial Cell Carcinoma; Urinary Bladder Disease; Urological Diseases
Keywords: Urothelial Cell Carcinoma; UCC; bladder cancer; vofatamab; FGFR3; invasive bladder cancer; targeted therapy; Transitional Cell Carcinoma; TCC; Phase 2; second line therapy; monoclonal antibody; docetaxel; combination therapy; Phase 1; monotherapy; B-701
MeSH Terms: conditions — Urinary Bladder Diseases; Urologic Diseases; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — vofatamab; B701 protein, Human herpesvirus 6; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vofatamab plus docetaxel (Active Comparator): IV infusion of docetaxel, 75 mg/m2, followed by IV infusion of vofatamab, 25 mg/kg, on day one of each 21-day cycle. One additional IV infusion of vofatamab (25 mg/kg) given on Day 8 of Cycle 1.
  Dosing with vofatamab and docetaxel will continue in each patient until disease progression, unacceptable toxicity, death, or study exit, including withdrawal of patient consent or study termination. Docetaxel treatment beyond 12 cycles of therapy may be considered at the discretion of the treating investigator and Medical Monitor.
  Interventions: Drug: Vofatamab; Drug: Docetaxel
- Placebo plus docetaxel (Placebo Comparator): IV infusion of docetaxel, 75 mg/m2, followed by IV infusion of placebo on day one of each 21-day cycle.
  One additional IV infusion of placebo given on Day 8 of Cycle 1. Dosing of docetaxel and placebo will continue in each patient until disease progression, unacceptable toxicity, death, or study exit, including withdrawal of patient consent or study termination. Docetaxel treatment beyond 12 cycles of therapy may be considered at the discretion of the treating investigator and Medical Monitor
  Interventions: Drug: Docetaxel; Drug: Placebo
- Vofatamab (Experimental): IV infusion vofatamab, 25 mg/kg on day one each 21-day cycle. One additional IV infusion of vofatamab (25 mg/kg) given on Day 8 of Cycle 1.
  Dosing of vofatamab will continue in each patient until disease progression, unacceptable toxicity, death, or study exit, including withdrawal of patient consent or study termination.
  Interventions: Drug: Vofatamab

INTERVENTIONS:
Drug: Vofatamab
  Other Names: B-701; MFGR1877S; R3Mab
  Arms: Vofatamab; Vofatamab plus docetaxel
Drug: Docetaxel
  Other Names: Docefrez; Taxotere
  Arms: Placebo plus docetaxel; Vofatamab plus docetaxel
Drug: Placebo
  Arms: Placebo plus docetaxel

SUMMARY:
This is a Phase 1/2(b), sequential, dose escalation, open-label, randomized expansion, multicenter, efficacy and safety study of vofatamab alone or in combination with docetaxel, or versus docetaxel in FGFR3 mutant/fusion subjects with Stage IV, locally advanced or metastatic UCC who have relapsed after, or are refractory to at least one prior line of chemotherapy. This study is divided into 3 phases: Phase 1b (Cohort 1), Phase 2 (Cohorts 2 and 3), and Phase 2b (Monotherapy Expansion Phase and Randomized Phase).

DETAILED DESCRIPTION:
This is a Phase 1/2(b), sequential, dose escalation, open-label, randomized expansion, multicenter, efficacy and safety study of vofatamab alone or in combination with docetaxel, or versus docetaxel in FGFR3 mutant/fusion subjects with Stage IV, locally advanced or metastatic UCC who have relapsed after, or are refractory to at least one prior line of chemotherapy. Vofatamab is a novel monoclonal antibody specific for fibroblast growth factor receptor 3 (FGFR3) that is being developed to target FGFR3-positive tumors.

This study is divided into 3 phases: Phase 1b (Cohort 1), Phase 2 (Cohorts 2 and 3), and Phase 2b (Monotherapy Expansion Phase and Randomized Phase).

ELIGIBILITY:
Key Disease Specific Inclusion Criteria:

1. Stage IV, locally advanced or metastatic (T4b, any N; or any T, N2-3) urothelial bladder cancer or TCC arising in another location of the urinary tract, including urethra, ureter, and renal pelvis
2. Histological or cytological diagnosis of UCC.
3. Relapsed after or are refractory to at least one prior line of chemotherapy which has not included a taxane (with the exception of Cohort 3 of Phase 2 and Phase 2b Monotherapy Expansion of Phase 2b which will allow the enrollment of patients with prior treatment with a taxane)
4. Subjects must have received at least one prior chemotherapeutic regimen (at least one cycle each) for advanced or metastatic/recurrent disease, of which at least one regimen included a platinum agent (unless contraindicated).
5. Prior neoadjuvant or adjuvant chemotherapy (without a taxane, except Cohort 3 of Phase 2 and Phase 2b Monotherapy Expansion, which will allow the enrollment of subjects with prior treatment with a taxane) is permitted and will not be counted as first-line chemotherapy, as long as the subject has not progressed within 12 months of the last dose.
6. Measurable disease according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

Phase 2 and Phase 2b Specific Inclusion Criteria:

1. Patient must be confirmed to have a FGFR3 genomic alteration at the time of documentation of advanced disease.
2. Relapsed after or are refractory to an immune checkpoint inhibitor. This inclusion criterion does not apply if the checkpoint inhibitor is contraindicated.

Main Exclusion Criteria:

* Prior anti-cancer therapy within 2 weeks prior to Cycle 1, Day 1
* Prior treatment with an inhibitor that is targeted primarily to FGFRs
* Clinically significant comorbid medical conditions or lab abnormalities
* History of major bleeding (requiring a blood transfusion ≥ 2 units) not related to a tumor within the past 12 months
* History of clinically significant coagulation or platelet disorder in the past 12 months
* Currently receiving anticoagulation treatment
* Incomplete healing from wounds from prior surgery
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection at screening
* Presence of positive test results for Hepatitis B or Hepatitis C
* Known history of human immunodeficiency virus (HIV) seropositive status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-06; Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainier Therapeutics, Study Chair — Rainier Therapeutics
Locations (49):
- United States (11):
  - Research Site, Gilbert, Arizona
  - Research Site, Goodyear, Arizona
  - Research Site, Duarte, California
  - Research Site, Miami, Florida
  - Reaserach Site, Fort Wayne, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Syracuse, New York
  - Research Site, Dallas, Texas
- Czechia (2):
  - Research Site, Olomouc
  - Research Site, Prague
- Italy (7):
  - Research Site, Ancona
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Negrar
  - Research Site, Siena
- South Korea (4):
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (9):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Valencia
  - Research Site, Vigo
- Research Site, Uppsala, Sweden
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (8):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Malatya
- United Kingdom (2):
  - Research Site, London
  - Research Site, Preston

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vofatamab Plus Docetaxel: IV infusion of docetaxel, 75 mg/m2, followed by IV infusion of vofatamab, 25 mg/kg, on day one of each 21-day cycle. One additional IV infusion of vofatamab (25 mg/kg) given on Day 8 of Cycle 1.
  Dosing with vofatamab and docetaxel will continue in each patient until disease progression, unacceptable toxicity, death, or study exit, including withdrawal of patient consent or study termination. Docetaxel treatment beyond 12 cycles of therapy may be considered at the discretion of the treating investigator and Medical Monitor.
  Vofatamab
  Docetaxel
- Vofatamab: IV infusion vofatamab, 25 mg/kg on day one each 21-day cycle. One additional IV infusion of vofatamab (25 mg/kg) given on Day 8 of Cycle 1.
  Dosing of vofatamab will continue in each patient until disease progression, unacceptable toxicity, death, or study exit, including withdrawal of patient consent or study termination.
  Vofatamab
- Placebo Plus Docetaxel: IV infusion of docetaxel, 75 mg/m2, followed by IV infusion of placebo on day one of each 21-day cycle.
  One additional IV infusion of placebo given on Day 8 of Cycle 1. Dosing of docetaxel and placebo will continue in each patient until disease progression, unacceptable toxicity, death, or study exit, including withdrawal of patient consent or study termination. Docetaxel treatment beyond 12 cycles of therapy may be considered at the discretion of the treating investigator and Medical Monitor
  Docetaxel
  Placebo
Period: Overall Study
Arm/Group | Vofatamab Plus Docetaxel | Vofatamab | Placebo Plus Docetaxel
Started | 41 | 30 | 0
Completed | 40 | 30 | 0
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in the placebo plus docetaxel group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vofatamab Plus Docetaxel | Vofatamab | Placebo Plus Docetaxel | Total
Number analyzed (Participants) | 40 | 30 | 0 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 12 | 0 | 32
  >=65 years | 20 | 18 | 0 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 0 | 13
  Male | 33 | 24 | 0 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 12 | 0 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 36 | 18 | 0 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Outcome: Progression Free Survival (PFS)
Description: Efficacy of vofatamab plus docetaxel, compared with docetaxel plus placebo, and vofatamab alone as measured by PFS; measured from randomization to first occurrence of disease progression (per RECIST v1.1) or death, whichever occurs first. A patient has had to receive at least one vofatamab dose. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 3-4 years
Measure: Mean (Standard Deviation); unit: Months
Groups:
- Mut/Fus Phase 1; Wild Type Phase 1; Mut/Fus Phase 2: Vofatamab plus Docetaxel
- Mut/Fus Phase 2 Monotherapy: Vofatamab Monotherpay
- Mut/Fus Phase 2b Monotherapy: Vofatamab Monotherapy
Arm/Group | Mut/Fus Phase 1 | Wild Type Phase 1 | Mut/Fus Phase 2 | Mut/Fus Phase 2 Monotherapy | Mut/Fus Phase 2b Monotherapy
Number analyzed (Participants) | 6 | 13 | 21 | 21 | 9
Months | 6.82 (5.35) | 2.83 (2.73) | 4.40 (4.15) | 4.45 (3.27) | 2.23 (1.45)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of informed consent through 30 days after the last dose of study drug.
Description: Safety was assessed through summaries of AEs, changes in key laboratory test results, ECGs and changes in vital signs.
Arm/Group | Vofatamab Plus Docetaxel | Vofatamab | Placebo Plus Docetaxel
All-Cause Mortality (participants affected / at risk) | 2/40 | 1/30 | 0/0
Serious Adverse Events (participants affected / at risk) | 21/40 | 6/30 | 0/0
Other Adverse Events (participants affected / at risk) | 40/40 | 30/30 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vofatamab Plus Docetaxel (N=40) | Vofatamab (N=30) | Placebo Plus Docetaxel (N=0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Pain (General disorders) | 2 (2) | 0 (0) | NA
Chills (General disorders) | 0 (0) | 1 (1) | NA
Fatigue (General disorders) | 1 (1) | 0 (0) | NA
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | NA
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | NA
Pyrexia (General disorders) | 1 (1) | 0 (0) | NA
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | NA
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | NA
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | NA
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | NA
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | NA
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | NA
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | NA
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | NA
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | NA
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | NA
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | NA
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | NA
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | NA
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | NA
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vofatamab Plus Docetaxel (N=40) | Vofatamab (N=30) | Placebo Plus Docetaxel (N=0)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 1 (1) | NA
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Abnormal ECG (Investigations) | 0 (0) | 1 (1) | NA
Absolute neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | NA
Ache (General disorders) | 1 (1) | 0 (0) | NA
Achilles tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | NA
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0) | NA
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Aerophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Airway compromise (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | NA
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 0 (0) | NA
ALP increased (Investigations) | 1 (1) | 0 (0) | NA
ALT increased (Investigations) | 4 (4) | 0 (0) | NA
Anemia (Blood and lymphatic system disorders) | 11 (11) | 2 (2) | NA
Anemia aggravated (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | NA
Ankle sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Anorexia (Metabolism and nutrition disorders) | 10 (10) | 2 (2) | NA
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | NA
Anxiety aggravated (Psychiatric disorders) | 1 (1) | 0 (0) | NA
Appetite lost (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | NA
Arthromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
AST increased (Investigations) | 4 (4) | 0 (0) | NA
Asthenia (General disorders) | 7 (7) | 0 (0) | NA
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1) | NA
Bilirubin total increased (Investigations) | 1 (1) | 0 (0) | NA
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | NA
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Bruising of foot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Burping (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | NA
Catheter leakage (Product Issues) | 1 (1) | 0 (0) | NA
Catheter occlusion (Product Issues) | 1 (1) | 0 (0) | NA
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | NA
Chest pain (General disorders) | 1 (1) | 0 (0) | NA
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | NA
Cold (Infections and infestations) | 1 (1) | 0 (0) | NA
Cold intolerance (General disorders) | 1 (1) | 0 (0) | NA
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Common cold (Infections and infestations) | 1 (1) | 0 (0) | NA
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | NA
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | NA
Constipation (Gastrointestinal disorders) | 11 (11) | 0 (0) | NA
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Contusion of foot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Costal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | NA
Cough aggravated (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | NA
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Cramp in hand (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Cramp legs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Creatinine increased (Investigations) | 7 (7) | 1 (1) | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Deep vein thrombosis leg (Vascular disorders) | 0 (0) | 1 (1) | NA
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | NA
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | NA
Desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Diarrhea (Gastrointestinal disorders) | 22 (22) | 2 (2) | NA
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | NA
Dorsal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Drug allergy (Immune system disorders) | 2 (2) | 0 (0) | NA
Drug fever (General disorders) | 1 (1) | 0 (0) | NA
Dysgeusia (Nervous system disorders) | 5 (5) | 0 (0) | NA
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | NA
Dyspnea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | NA
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Dysuria aggravated (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Edema legs (General disorders) | 2 (2) | 0 (0) | NA
Edema of lower extremities (General disorders) | 4 (4) | 0 (0) | NA
Edematous feet (General disorders) | 1 (1) | 0 (0) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | NA
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Erythema facial (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Eye redness (Eye disorders) | 1 (1) | 0 (0) | NA
Eyes tearing (Eye disorders) | 1 (1) | 0 (0) | NA
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Fatigue (General disorders) | 17 (17) | 0 (0) | NA
Fatigue aggravated (General disorders) | 3 (3) | 0 (0) | NA
Febrile reaction (General disorders) | 1 (1) | 0 (0) | NA
Fecal incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0) | NA
Fever (General disorders) | 19 (19) | 1 (1) | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | NA
Flashing lights (Eye disorders) | 1 (1) | 0 (0) | NA
Flu like symptoms (General disorders) | 2 (2) | 0 (0) | NA
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Flushed face (Vascular disorders) | 2 (2) | 0 (0) | NA
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Fractured ribs (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Gas pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Gastralgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
General body pain (General disorders) | 0 (0) | 1 (1) | NA
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
GGT increased (Investigations) | 1 (1) | 0 (0) | NA
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Hair loss (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | NA
Headache (Nervous system disorders) | 4 (4) | 0 (0) | NA
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Hematuria (Renal and urinary disorders) | 3 (3) | 1 (1) | NA
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | NA
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | NA
Hypercalcemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | NA
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | NA
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Hyperpyrexia (General disorders) | 0 (0) | 1 (1) | NA
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | NA
Hypertension aggravated (Vascular disorders) | 1 (1) | 0 (0) | NA
Hypertension worsened (Vascular disorders) | 1 (1) | 0 (0) | NA
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | NA
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | NA
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | NA
Hyponatremia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | NA
Hyporexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | NA
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | NA
Iliac vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | NA
Inappetence (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Inferior venacaval thrombosis (Vascular disorders) | 0 (0) | 1 (1) | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | NA
Infusion site erythema (General disorders) | 1 (1) | 0 (0) | NA
Infusion site redness (General disorders) | 1 (1) | 0 (0) | NA
Insomnia (Psychiatric disorders) | 6 (6) | 1 (1) | NA
Intermittent fever (General disorders) | 1 (1) | 0 (0) | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Itch (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Itching eyes (Eye disorders) | 1 (1) | 0 (0) | NA
Itchy throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Joint ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Leg pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | NA
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | NA
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | NA
Lipase increased (Investigations) | 1 (1) | 0 (0) | NA
Localized itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | NA
Loose stools (Gastrointestinal disorders) | 3 (3) | 0 (0) | NA
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | NA
Low back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | NA
Lower extremities weakness of (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | NA
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | NA
Lymphocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | NA
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Malaise (General disorders) | 1 (1) | 0 (0) | NA
Malleolus edema (General disorders) | 1 (1) | 0 (0) | NA
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | NA
Mucositis (General disorders) | 6 (6) | 0 (0) | NA
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Muscular pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | NA
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | NA
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Nasal sinus discharge (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Nausea (Gastrointestinal disorders) | 15 (15) | 2 (2) | NA
Nausea aggravated (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Neurogenic claudication (Nervous system disorders) | 1 (1) | 0 (0) | NA
Neuropathic pain (Nervous system disorders) | 1 (1) | 0 (0) | NA
Neuropathy (Nervous system disorders) | 4 (4) | 0 (0) | NA
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0) | NA
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0) | NA
Neutrophil count decreased (Investigations) | 5 (5) | 0 (0) | NA
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | NA
Nightmares (Psychiatric disorders) | 1 (1) | 0 (0) | NA
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | NA
Numbness in feet (Nervous system disorders) | 1 (1) | 0 (0) | NA
Onychodystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | NA
Oral ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | NA
Orthostatic dizziness (Nervous system disorders) | 1 (1) | 0 (0) | NA
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | NA
Pain abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Pain aggravated (General disorders) | 1 (1) | 0 (0) | NA
Pain flank (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Pain in thigh (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | NA
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | NA
Penile bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | NA
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | NA
Phlebitis (Vascular disorders) | 2 (2) | 0 (0) | NA
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | NA
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | NA
Postoperative pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Protein total increased (Investigations) | 1 (1) | 0 (0) | NA
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | NA
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | NA
Puncture wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
QT prolonged (Investigations) | 1 (1) | 0 (0) | NA
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | NA
Rash both legs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Rash face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
Redness of face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Right arm paresis (Nervous system disorders) | 1 (1) | 0 (0) | NA
Right cataract (Eye disorders) | 1 (1) | 0 (0) | NA
Right lower quadrant pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Rigors (General disorders) | 1 (1) | 0 (0) | NA
Ringing in ears (Ear and labyrinth disorders) | 1 (1) | 0 (0) | NA
Sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | NA
SGOT increased (Investigations) | 1 (1) | 0 (0) | NA
Shivers (General disorders) | 1 (1) | 0 (0) | NA
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | NA
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | NA
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | NA
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
Skin peeling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | NA
Skin ulcer bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA
Sleeplessness (Psychiatric disorders) | 1 (1) | 0 (0) | NA
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | NA
Sores mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Spinal stenosis NOS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Sputum bloody (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
ST segment elevation (Investigations) | 1 (1) | 0 (0) | NA
Stomach cramps (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Stomachache (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Stye (Infections and infestations) | 1 (1) | 0 (0) | NA
Swelling abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Swelling of legs (General disorders) | 1 (1) | 0 (0) | NA
Swollen joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Swollen thumb (General disorders) | 1 (1) | 0 (0) | NA
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | NA
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | NA
Tearing eyes (Eye disorders) | 1 (1) | 0 (0) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA
Tingling (Nervous system disorders) | 1 (1) | 0 (0) | NA
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Upper abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Upper limb edema (General disorders) | 1 (1) | 0 (0) | NA
Upper respiratory infection (Infections and infestations) | 5 (5) | 0 (0) | NA
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | NA
Urethral discharge (Renal and urinary disorders) | 0 (0) | 1 (1) | NA
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | NA
Urinary infection (Infections and infestations) | 0 (0) | 1 (1) | NA
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0) | NA
Urinary tract infection (Infections and infestations) | 6 (6) | 0 (0) | NA
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | NA
UTI (Infections and infestations) | 1 (1) | 0 (0) | NA
Vaginal yeast infection (Infections and infestations) | 1 (1) | 0 (0) | NA
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | NA
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (3) | NA
WBC decreased (Investigations) | 1 (1) | 0 (0) | NA
Weakness (General disorders) | 2 (2) | 0 (0) | NA
Weakness generalized (General disorders) | 2 (2) | 0 (0) | NA
Weight loss (Investigations) | 1 (1) | 0 (0) | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Wheezing aggravated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | NA
Xerophthalmia (Eye disorders) | 2 (2) | 0 (0) | NA
Xerostomia (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA
Zona (Infections and infestations) | 1 (1) | 0 (0) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT02401542/Prot_SAP_000.pdf